CLINICAL TRIAL: NCT06186180
Title: Effects of Inspiratory Muscle Training on Diaphragm Thickness, Inspiratory Muscle Strength and Non-especific Shoulder Pain in Federated Tennis Player
Brief Title: Inspiratory Muscle Training on Diaphragm Thickness, Inspiratory Muscle Strength and Shoulder Pain in Tennis Player
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 46/2022
Record Dates: First submitted 2023-12-08; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Pain; Inspiratory Muscle Training
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Single blinded randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inspiratory muscle training (Experimental): They will perform 5 sets of 10 repetitions with a 1-minute rest between sets, 5 days a week, using a specific respiratory muscle training device.
  Interventions: Other: inspiratory muscle training
- control (No Intervention): no intervention

INTERVENTIONS:
Other: inspiratory muscle training — They will perform 5 sets of 10 repetitions with a 1-minute rest between sets, 5 days a week, using a specific respiratory muscle training device
  Arms: inspiratory muscle training

SUMMARY:
Shoulder pain is one of the most common musculoskeletal conditions among athletes and sports enthusiasts who engage in overhead sports, and it can be highly disabling. Since the shoulder is one of the joints with the greatest range of motion in the human body, it is important to seek strategies that address trunk stability comprehensively to achieve full and effective joint mobility. The central role of the diaphragm in trunk stabilization has been the subject of research for over 50 years, although the exact mechanisms are still not fully understood.

The objective of this study is to assess the effects of inspiratory muscle training on diaphragm thickness, inspiratory muscle strength, and shoulder pain in adult tennis players with non-specific shoulder pain.

This is a single-blind, randomized controlled clinical trial. The intervention will last for 8 weeks. Patients with non-specific shoulder pain will be randomly assigned to one of two groups. The experimental group will undergo specific inspiratory muscle training, while the control group will receive no specific training intervention. Measurements of diaphragm thickness, inspiratory muscle strength, and shoulder pain will be taken before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* tennis player who suffered from inespecific shoulder pain
* training at least two times per week
* Have experienced at least 1 episode of non-specific shoulder pain in the last month
* A positive result on diagnostic tests performed: Neer Test and Jobe Test

Exclusion Criteria:

* Having taken anti-inflammatories or muscle relaxants within the last 72 hours before the study
* pregnancy
* Previous diagnosis of respiratory or neurological diseases
* Previous surgeries, fractures, and dislocations in the dominant shoulder
* Inability to follow instructions during the study
* All those for whom measuring maximum inspiratory pressure is contraindicated: unstable angina, recent myocardial infarction (within 4 weeks of the event) or myocarditis, uncontrolled systemic hypertension, recent pneumothorax, post-lung biopsy surgery of less than one week, postoperative abdominal or genitourinary surgery of less than 6 months, and urinary incontinence

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
diaphragm thickness | before and after the 8 weeks of inspiratory muscle training
  The thickness of the diaphragm will be measured using ultrasound, with a Toshiba Xario 100 ultrasound machine. Image acquisition will be performed by a physiotherapist experienced in musculoskeletal ultrasound. A linear probe (Toshiba PLT-805AT) with a frequency range of 8 to 12 MHz and a 54 mm probe footprint will be used to perform transcostal measurements at rest and in the supine position, using the B-Mode of ultrasound imaging (preset at 3 cm depth, 12MHz frequency, 64 gain points, 64 dynamic range points, and a single focus point located at 2 cm depth). Bilateral transcostal images will be obtained with the linear probe placed perpendicular to the last intercostal space, allowing for adequate visualization of the diaphragm without invasion of lung tissue during normal breathing

SECONDARY OUTCOMES:
maximal inspiratory pressure | before and after the 8 weeks of inspiratory muscle training
  Inspiratory muscle strength will be measured using a portable device, POWERbreathe KH1. It is a simple test in which the subject performs a maximal forced inspiration against an airway occlusion mechanism in the mouth after a slow and prolonged near-residual volume expiration, yielding the maximum inspiratory pressure (MIP) value. The evaluation will be conducted with the subject seated in a chair (knees and hips at 90º), and their nose will be occluded with a clip. The advantage of this test is that it provides a quick and non-invasive way to assess inspiratory muscle strength through maximum inspiratory pressure. Three measurements will be taken, with 1 minute of rest between each measurement, and the best of the three will be selected, provided that there is no more than a 10% difference between them
shoulder pain through VAS | before and after the 8 weeks of inspiratory muscle training
  Shoulder pain will be measured using the Visual Analog Scale for Pain (VAS), which is a valid and reliable measure for assessing pain. Its validity has been demonstrated with high correlations to other pain measures (r=0.62 to 0.91), and it has good test-retest reliability (r=0.94 to 0.71)(31). Participants will indicate their maximum pain sensation during the past week using a 100-mm VAS, where 0 represents 'no pain' and 100 represents 'extreme and unbearable pain
Upper trapezius, levator scapulae and middle deltoid pain pressure threshold | before and after the 8 weeks of inspiratory muscle training
  the measurement of pressure pain using an algometer will be performed at the upper trapezius, the levator scapulae, and the middle deltoid, as shown by studies at the shoulder level. The contact area will be 10mm, and it will be applied at a rate of 30 kPa/s. Patients will be instructed to signal the moment they feel the first sensation of pain
The Shortened Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) | before and after the 8 weeks of inspiratory muscle training
  The Shortened Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) consists of 11 questions that assess daily activities, symptoms, social function, work function, sleep, and confidence. There are 5 points, with 1 indicating no difficulty and 5 indicating impossibility. The score is converted to a 100-point scale, with 100 representing the highest level of disability

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Davinia Vicente-Campos, Pozuelo de Alarcón, Madrid
  - Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid

IPD SHARING:
Plan to Share IPD: No